CLINICAL TRIAL: NCT00480181
Title: A Comparative, Single Center, Randomized, Double-blinded, Parallel, Placebo-controlled Study to Evaluate the Efficacy of Nabilone (Cesamet) as Adjunctive Therapy to Gabapentin (Neurontin) in the Management of Neuropathic Pain (NPP) Symptoms in Subjects With Multiple Sclerosis (MS)
Brief Title: Efficacy and Safety Evaluation of Nabilone as Adjunctive Therapy to Gabapentin for the Management of Neuropathic Pain in Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Dr. M. Namaka, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2007:051
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2011-03

CONDITIONS: Neuropathic Pain; Multiple Sclerosis
Keywords: Neuropathic pain; Multiple Sclerosis; Nabilone; Gabapentin
MeSH Terms: conditions — Neuralgia; Multiple Sclerosis | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: nabilone
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: nabilone — Cesamet (nabilone) capsules given at titrating dosages as per protocol.
  Other Names: Cesamet
  Arms: Active
Other: placebo — placebo capsules (identical appearance to Cesamet) given at titrating dosages as per protocol.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether nabilone (Cesamet) when used as an adjunctive agent with gabapentin (Neurontin) provides significantly improved pain relief over gabapentin alone for the management of neuropathic pain in MS.

DETAILED DESCRIPTION:
Neuropathic pain syndromes, which occur due to damage to central and/or peripheral nerve axons, are often more difficult to manage and are commonly refractory to the conventional analgesia approach described by the World Health Organization, including NSAIDs and narcotic agents. These pain syndromes are often described by symptoms of burning, stabbing, crawling, shock-like, numbness and/or tingling, and can be quite concerning to the patient, especially when there is an inadequate response to treatment. It has been estimated that the prevalence of chronic pain in MS ranges anywhere from 30-90%, placing it as the second worst disease-induced symptom experienced by this patient population.

The pathophysiologic causes of this pain syndrome are complex and multifaceted, with no one specific link attributed to the pain response. Due to the complexity of neuropathic pain - which is only partially understood at best - it may be necessary in many cases to treat the source of the pain with more than one agent in order to address the many different contributors to this pain process. More thorough review of how the currently available agents for NPP work together would provide clinicians with safety and efficacy data which would aid in providing optimal pain management.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-65 years old with clinically definite RRMS
* EDSS of < 6.5
* Current treatment with gabapentin that is not effective at a stabilized dose of (>1800mg/day) for at least 1 month.
* Visual Analogue Scale score for NPP symptoms > 5; pain present for at least 3 months
* Negative serum pregnancy test for all females of childbearing age; not currently breastfeeding
* No history of alcohol or substance abuse
* No history of non-psychotic emotional disorders
* No significant hepatic or renal insufficiency
* No significant cardiovascular disease or hypertension
* No known hypersensitivity and/or allergy to nabilone or its derivatives
* No current use of cannabinoid or related products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
VAS | 9 weeks

SECONDARY OUTCOMES:
SF MPQ | 9 weeks
SF-36 | 9 weeks
PGIC | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Namaka, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Multiple Sclerosis Clinic, Winnipeg, Manitoba, Canada